CLINICAL TRIAL: NCT04363879
Title: Comparing Two Types of Endometrial Activation Prior to Embryo Transfer: A Pilot Study
Brief Title: Comparing Two Types of Endometrial Activation Prior to Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-14-06B
Record Dates: First submitted 2020-04-22; First posted 2020-04-27 (Actual); Results first posted 2020-05-27 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Infertility; Endometrial Disorder
Keywords: Endometrial scratch
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Parallel treatment arms for two types of endometrial scratch
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometrial scratch with Pipelle curette (Active Comparator): For patients in the Pipelle curette group, physicians inserted the Pipelle curette into the uterus and removed an adequate endometrial sample using vigorous motion.
  Interventions: Procedure: Endometrial scratch with Pipelle curette
- Endometrial scratch with Shepard catheter (Experimental): For patients in the Shepard catheter group, physicians performed a four-quadrant scratch technique by inserting the Shepard insemination catheter into the uterus at 12:00. The catheter was then turned one-quarter turn and withdrawn. This was repeated two more times so that four endometrial quadrants were touched by the catheter at 12:00, 3:00, 6:00, and 9:00.
  Interventions: Procedure: Endometrial scratch with Shepard catheter

INTERVENTIONS:
Procedure: Endometrial scratch with Pipelle curette — For patients in the Pipelle curette group, physicians inserted the Pipelle curette into the uterus and removed an adequate endometrial sample using vigorous motion.
  Other Names: Endometrial activation, endometrial injury
  Arms: Endometrial scratch with Pipelle curette
Procedure: Endometrial scratch with Shepard catheter — For patients in the Shepard catheter group, physicians performed a four-quadrant scratch technique by inserting the Shepard insemination catheter into the uterus at 12:00. The catheter was then turned one-quarter turn and withdrawn. This was repeated two more times so that four endometrial quadrants were touched by the catheter at 12:00, 3:00, 6:00, and 9:00.
  Other Names: Endometrial activation, endometrial injury
  Arms: Endometrial scratch with Shepard catheter

SUMMARY:
To determine if two types of endometrial activation (Pipelle curette or Shepard catheter) prior to embryo transfer result in similar live birth rates. Also to determine if patients experience similar pain from both types of endometrial activation.

DETAILED DESCRIPTION:
Assisted reproductive technologies (ART), including in vitro fertilization (IVF), are methods used to treat infertility, which affects approximately 10% reproductive aged women. Physicians at the Women's Institute perform over 300 embryo transfer procedures every year. Despite advances and improvements in ART over the past three decades, clinical pregnancy rate and live birth rate remain 30-40% and 20-30%. Implantation is essential for successful ART and IVF procedures, and many interventions have been studied to possibly improve implantation rates and thus pregnancy and live birth rates.

Endometrial activation is one such intervention, sometimes referred to as endometrial "activation" or "scratch," and it is defined as "intentional endometrial injury, such as endometrial biopsy or curettage, in women undergoing ART".

A previous study found that implantation rates, clinical pregnancy rates, and live birth rates were more than twofold higher in women who underwent endometrial biopsy in the cycle before subsequent IVF treatment. Another study which examines endometrial activation prior to IVF similarly has concluded that endometrial activation prior to the embryo transfer cycle significantly improves clinical pregnancy rates and live birth rates in women undergoing ART. Although the type of endometrial procedure is not specified, the timing activation was found be most effective when performed in the cycle prior to the embryo transfer.

The mechanism of increase endometrial receptivity is still unknown; however three proposed hypothesis exist. The first hypothesis proposes that local activation of the endometrium induces endometrial decidualization which increases the probability of embryo implantation. The second hypothesis is that endometrial healing following endometrial activation increases secreted cytokines, interleukins, growth factors, macrophages, and dendritic cells which are beneficial to embryo implantation. The final hypothesis suggests that endometrial maturation is abnormally advanced during ovarian stimulation, so endometrial activation may lead to better synchronicity between the endometrium and the embryo..

Endometrial activation has been found to have clear benefit in pregnancy and live birth rates in a previous study, however no uniform technique has been determined. The objective of this study is to compare two types of endometrial disruption - a vigorous endometrial biopsy with a Pipelle curette and a four quadrant endometrial "scratch" using a Shepard insemination catheter - to determine if the live birth rates are equivalent for the two methods. The investigators also will compare pain with the two types of endometrial activation. By comparing two distinct types of endometrial activation, the goal is to determine which method is both effective and tolerable to patients.

The Shepherd catheter is a 1.8 mm malleable insemination catheter that can be curved to traverse the cervix. It is also used by some physicians in the Women's Institute to perform saline infusion sonography. When the catheter is inserted under ultrasound guidance, it is often placed in the subendometrial tissue, and causes deflection and disruption of the endometrium but is tolerated well. The Pipelle is a 3.1 mm semi-rigid catheter with an internal stylet plunger. A biopsy is performed by placing the catheter into the uterus, withdrawing the stylet to create suction, and aspirating endometrial tissue into the catheter.

A study done by Leclair et al. found that the mean pain that women had when the Pipelle was used for an endometrial biopsy was 6.2±2.4 on a visual analog scale from 1-10 (5). Pain with the Shepard catheter has not been studied when it is used for endometrial biopsy.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing embryo transfer who are in the cycle prior to their embryo transfer

Exclusion Criteria:

* Patients not undergoing embryo transfer
* Known pregnancy
* Active pelvic infection
* Known endometrial hyperplasia or cancer
* Inability to tolerate endometrial catheter placement
* Severe cervical stenosis
* Patients who will receive operative hysteroscopy in the cycle prior to embryo transfer

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Hurst, MD, Principal Investigator — Wake Forest University Health Sciences; Kathryn Goldrick, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual patient data with other researchers.

REFERENCES:
- [Background] Nastri CO, Ferriani RA, Raine-Fenning N, Martins WP. Endometrial scratching performed in the non-transfer cycle and outcome of assisted reproduction: a randomized controlled trial. Ultrasound Obstet Gynecol. 2013 Oct;42(4):375-82. doi: 10.1002/uog.12539. Epub 2013 Sep 2. PMID 23754314
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Background] Nastri CO, Lensen SF, Gibreel A, Raine-Fenning N, Ferriani RA, Bhattacharya S, Martins WP. Endometrial injury in women undergoing assisted reproductive techniques. Cochrane Database Syst Rev. 2015 Mar 22;(3):CD009517. doi: 10.1002/14651858.CD009517.pub3. PMID 25803542
- [Background] Leclair CM, Zia JK, Doom CM, Morgan TK, Edelman AB. Pain experienced using two different methods of endometrial biopsy: a randomized controlled trial. Obstet Gynecol. 2011 Mar;117(3):636-641. doi: 10.1097/AOG.0b013e31820ad45b. PMID 21343767
- [Background] Nastri CO, Gibreel A, Raine-Fenning N, Maheshwari A, Ferriani RA, Bhattacharya S, Martins WP. Endometrial injury in women undergoing assisted reproductive techniques. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD009517. doi: 10.1002/14651858.CD009517.pub2. PMID 22786529

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endometrial Scratch With Pipelle Curette | Endometrial Scratch With Shepard Catheter
Started | 78 | 92
Completed | 78 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Scratch With Pipelle Curette | Endometrial Scratch With Shepard Catheter | Total
Number analyzed (Participants) | 78 | 92 | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (4.6) | 34.2 (3.9) | 34.0 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 92 | 170
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 75 | 91
  Unknown or Not Reported | 62 | 17 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 78 | 92 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Live Births Per Transfers Performed
Description: Number (count) of births per number of subjects undergoing embryo transfer
Time Frame: Collected up to 1 year after the last embryo transfer
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Scratch With Pipelle Curette | Endometrial Scratch With Shepard Catheter
Number analyzed (Participants) | 78 | 92
Participants | 37 | 43

2. Secondary Outcome: Pain Quantifcation After Endometrial Scratch
Description: Pain assessed by Visual analog scale (Numeric rating scale, units from 1-10 with 1 being no pain and 10 being maximum pain)
Time Frame: Immediately following endometrial scratch
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Endometrial Scratch With Pipelle Curette | Endometrial Scratch With Shepard Catheter
Number analyzed (Participants) | 78 | 92
score on a scale | 3.9 (2.2) | 3.0 (2.4)

3. Secondary Outcome: Number (Count) of Positive Pregnancy Tests Per Number of Subjects Undergoing Embryo Transfer
Time Frame: Collected up to 1 year after the last embryo transfer
Measure: Number; unit: positive pregnancy tests
Arm/Group | Endometrial Scratch With Pipelle Curette | Endometrial Scratch With Shepard Catheter
Number analyzed (Participants) | 78 | 92
positive pregnancy tests | 56 | 62

4. Secondary Outcome: Number (Count) of Pregnancies Per Number of Patients Undergoing Embryo Transfer
Time Frame: Collected up to 1 year after the last embryo transfer
Measure: Number; unit: number of pregnancies
Arm/Group | Endometrial Scratch With Pipelle Curette | Endometrial Scratch With Shepard Catheter
Number analyzed (Participants) | 78 | 92
number of pregnancies | 44 | 55

ADVERSE EVENTS:
Time Frame: From start of study until 1 year after last embryo transfer
Description: There were no adverse events
Arm/Group | Endometrial Scratch With Pipelle Curette | Endometrial Scratch With Shepard Catheter
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/92
Other Adverse Events (participants affected / at risk) | 0/78 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT04363879/Prot_SAP_000.pdf